CLINICAL TRIAL: NCT06929416
Title: Relationship Between Serum Estrogen Concentration and Propofol Injection Pain: A Prospective and Observational Study
Brief Title: Estrogen and Propofol Injection Pain
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Mahmut Sami TUTAR, Associate Professor, Department of Anesthesiology and Reanimation, Konya City Hospital
Other Study IDs: 2.02.2025-35906
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Pain; Estradiol; Assisted Reproductive Techniques
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Women Undergoing IVF With Supraphysiological Estrogen Levels
- 2: Women Undergoing Elective Surgery With Normal Estrogen Levels

SUMMARY:
This prospective observational study investigates the relationship between serum estrogen concentration and the incidence and severity of propofol injection pain (PIP) in female patients undergoing general anesthesia. The study will include 90 ASA I-II female patients aged 18-45. One group will consist of IVF patients with elevated estrogen levels, while the control group will include patients with normal estrogen levels undergoing other elective procedures. Pain will be assessed using a standardized four-point behavioral pain scale. The findings may enhance understanding of hormonal influences on pain and contribute to improving patient comfort during anesthesia induction.

DETAILED DESCRIPTION:
This prospective observational study aims to evaluate the association between serum estrogen levels and the incidence and severity of propofol injection pain (PIP) in adult female patients undergoing general anesthesia. Although propofol is a widely used intravenous anesthetic, it frequently causes pain upon injection. Estrogen is believed to play a role in modulating pain perception and inflammatory responses, yet the effects of elevated estrogen levels on PIP are not well understood.

The study will be conducted at a single tertiary hospital and will include 90 ASA I-II female patients aged 18-45 years. One group will consist of IVF patients with elevated serum estradiol levels due to controlled ovarian stimulation. The control group will include patients with normal estradiol levels scheduled for elective procedures under general anesthesia. Preoperative serum estradiol levels will be recorded, and injection pain will be evaluated using a validated four-point behavioral pain scale based on vocal response, facial expression, limb movement, and tearfulness.

Anesthesia induction will follow standard clinical practice without additional interventions. Pain data will be collected through routine clinical observation. The results may offer new insights into hormonal modulation of acute nociceptive responses and help improve patient experiences during anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18 and 45 years
* American Society of Anesthesiologists (ASA) physical status I or II
* Scheduled for surgery under general anesthesia
* Availability of a preoperative serum estradiol (E2) level
* For Group 1: Undergoing IVF procedure with supraphysiological E2 levels (>350 pg/mL)
* For Group 2: Undergoing elective surgery with normal E2 levels (15-350 pg/mL)

Exclusion Criteria:

* ASA physical status III or IV
* Pregnant patients
* Perimenopausal women
* Male patients
* Patients younger than 18 or older than 45 years
* History of psychiatric disorders
* Patients undergoing emergency surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of adult female patients aged 18 to 45 years, with ASA physical status I or II, who are scheduled for elective surgical procedures under general anesthesia. Participants will be divided into two groups based on their preoperative serum estradiol levels: one group will include women undergoing IVF procedures with supraphysiological estrogen levels, and the other will consist of patients with normal estrogen levels undergoing unrelated elective surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Propofol Injection Pain | Immediately during induction of anesthesia
  Presence or absence of pain during propofol injection, assessed through patient response (verbal reaction, facial grimacing, arm withdrawal, or tearing) and/or verbal confirmation during anesthesia induction. Comparison between patients with normal and supraphysiological estradiol levels.

SECONDARY OUTCOMES:
Severity of Propofol Injection Pain | Immediately during induction of anesthesia
  Pain intensity during propofol injection will be graded using a validated 4-point behavioral scale:
  0 = no pain,
  1. = mild pain (reported only when asked, without behavioral signs),
  2. = moderate pain (reported when asked and with behavioral signs),
  3. = severe pain (spontaneous report with strong vocal, facial, or physical reactions such as tearing).
Postoperative Injection Site Reactions | Within 24 hours after surgery
  Presence of local signs such as redness, swelling, tenderness, or edema at the injection site will be assessed by a blinded anesthesiologist within 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Tutar, MD, Study Chair — KONYA CITY HOSPİTAL
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy considerations and lack of prior consent for data sharing.